CLINICAL TRIAL: NCT00224653
Title: Comparison Between Volume Controlled Ventilation and Pressure Controlled Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P040405; PS040405
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2006-04-13 (Estimated); Status verified 2005-09

CONDITIONS: Obesity; Reduced Lung Compliance.; Anesthesia.; Laparoscopy.
Keywords: Obesity.; Respiration. Respiration, artificial.; Ventilation. Pressure controlled. Volume controlled.
MeSH Terms: conditions — Obesity | interventions — Respiration, Artificial

INTERVENTIONS:
Procedure: Mechanical Ventilation

SUMMARY:
To assess the potential benefits on mechanical ventilation plateau pressure of pressure controlled mode versus volume controlled mode for laparoscopic bariatric surgery in obese patients (BMI > 35). High plateau pressures encountered in obese patients due to their reduced pulmonary compliance could be lowered using pressure controlled mechanical ventilation.

DETAILED DESCRIPTION:
All patients are over 18 years old and give their inform consent after approval of the study protocol by an ethic committee. Anesthesia is standardized and all patients are intubated. Precise protocols are used to perform pressure and volume controlled ventilation in order to regulate End-Tidal CO2 between 33 and 35 mmHg. Primary goal is comparison of plateau pressures observed in the 2 ventilation modes after 45 minutes of pneumoperitoneum. Secondary goals are : comparison of PaO2 and PaCO2 after 45 minutes of pneumoperitoneum and after 2 hours spent in post-anesthesia care unit ; comparison of total respiratory resistances and peak flow generated between the 2 modes.

ELIGIBILITY:
Inclusion Criteria:

* patients are over 18 years old and give their inform consent
* morbid obesity(BMI>35)
* laparoscopic bariatric surgery

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-01; Study Completion 2005-06

PRIMARY OUTCOMES:
Plateau pressures generated by mechanical ventilation after 45 minutes of pneumoperitoneum.

SECONDARY OUTCOMES:
Comparison of PaO2 and PaCO2 after 45 minutes of pneumoperitoneum and after 2 hours spent in post-anesthesia care unit ; comparison of total respiratory resistances and peak flow generated between the 2 modes.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CADI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Georges Pompidou European Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Frappier J, Guenoun T, Journois D, Philippe H, Aka E, Cadi P, Silleran-Chassany J, Safran D. Airway management using the intubating laryngeal mask airway for the morbidly obese patient. Anesth Analg. 2003 May;96(5):1510-1515. doi: 10.1213/01.ANE.0000057003.91393.3C. PMID 12707159